CLINICAL TRIAL: NCT03298347
Title: Caffeine for Preterm Infants With Apnea of Prematurity(AOP): a Randomized Controlled Trial
Brief Title: Caffeine for Preterm Infants With Apnea of Prematurity(AOP)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Ma Juan, Director, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201733
Record Dates: First submitted 2017-09-27; First posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Caffeine; Apnea of Prematurity
MeSH Terms: conditions — Apnea | interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 80mg/kg of caffeine (Experimental): 80mg/kg of caffeine is given to treat AOP.
  Interventions: Drug: 80mg/kg of caffeine
- 20mg/kg of caffeine (Active Comparator): 20mg/kg of caffeine is given to treat AOP.
  Interventions: Drug: 20mg/kg of caffeine

INTERVENTIONS:
Drug: 80mg/kg of caffeine — 80mg/kg of caffeine is given to treat AOP
  Arms: 80mg/kg of caffeine
Drug: 20mg/kg of caffeine — 20mg/kg of caffeine is given to treat AOP
  Arms: 20mg/kg of caffeine

SUMMARY:
Nowadays,caffein is commonly used for AOP, and it reduces the intubation rate in preterm infants. However, intubation is needed in about 20%-50% of partial neonates. How to reduce the intubation rate effectively is a challenge for neonatologists.

DETAILED DESCRIPTION:
Less evidences about more dose of caffein used in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* gestational age less than 32 weeks;
* appear AOP;
* parents'consents are obtained.

Exclusion Criteria:

* major congenital abnormalities;
* Parents' rejection

Ages: 1 Minute to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
the rate of AOP | within 100 days
  AOP appears again in preterm infants

CONTACTS AND LOCATIONS:
Overall Officials: Shi Yuan, MD;PhD, Study Director — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (1):
- Daping Hospital and the Research Institute of Surgery of the Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided